CLINICAL TRIAL: NCT01431508
Title: An Open-label, Single Arm, Prospective Study to Evaluate the Safety and Anti-hypertensive Efficacy of Losartan 50 mg / Hydrochlorothiazide (HCTZ) 12.5 mg Combination in Patients With Mild to Moderate Essential Hypertension
Brief Title: A Study of Safety and Efficacy in MK-0954A Combination in Participants With Hypertension (MK-0954A-373 AM3)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0954A-373
Record Dates: First submitted 2011-09-07; First posted 2011-09-09 (Estimated); Results first posted 2011-11-22 (Estimated); Last update posted 2024-05-22 (Actual); Status verified 2022-02

CONDITIONS: Hypertension
Keywords: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Losartan; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Losartan 50 mg / HCTZ 12.5 mg (Experimental): Participants with mild to moderate essential hypertension who will receive Losartan 50 mg / HCTZ 12.5 mg once-a-day for 12 weeks.
  Interventions: Drug: Losartan 50 mg / HCTZ 12.5 mg

INTERVENTIONS:
Drug: Losartan 50 mg / HCTZ 12.5 mg — Losartan 50 mg / HCTZ 12.5 mg tablet once daily for 12 weeks
  Other Names: MK-0954A

SUMMARY:
This study is being conducted to evaluate the safety and antihypertensive efficacy of MK-0954A (Losartan 50 mg / Hydrochlorothiazide (HCTZ) 12.5 mg) in participants with mild to moderate essential hypertension.

ELIGIBILITY:
Inclusion criteria:

* Participant will have reached the legal age by the time of entrance into the run-in period.
* Participant has no active medical problem, other than essential hypertension,

which might of itself or by this treatment significantly affect the Participant's blood pressure.

- Participants diagnosed with mild to moderate essential hypertension or

hypertension accompanying with established cardiovascular (CV) and renal diseases who are receiving antihypertensive regimen (exclude diuretic), yet not attaining to treatment goal*.

* Note: For essential hypertension, the goal is to reduce the blood pressure to less than 140/90. For hypertension with established CV and renal diseases, the BP goal is < 130/80. (According to 2007 European Society of Hypertension (ESH) - European Society of Cardiology (ESC) guideline)

* Participant is either receiving antihypertensive therapy or no treatment.
* Participants with stable diabetes mellitus may enter the study.

Exclusion criteria:

* Pregnant or lactating females.
* Secondary hypertension of any etiology (such as unilateral or bilateral renal

disease, renal artery stenosis, coarctation of the aorta, pheochromocytoma).

* History of malignant hypertension.
* Sitting systolic blood pressure >210 mmHg at Visit 1 (Day 0).
* Participants with unresolved cerebrovascular accident or transient ischemic attack in the acute stage at visit 1.
* A clinically confirmed myocardial infarction within the recent 3 months.
* Angina pectoris.
* Clinically important cardiac arrhythmia.
* History of unexplained syncope within the prior 2 years, or a known syncopal

disorder.

- Presence of hemodynamically significant obstructive valvular disease of

cardiomyopathy.

* Percutaneous coronary angioplasty or coronary artery bypass surgery within the prior 3 months of visit 1.
* Participant with a single functioning kidney.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-08-01 (Actual); Primary Completion 2009-06-01 (Actual); Study Completion 2009-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Du-Yi Lee, M.D., Principal Investigator — Cheng Ching General Hospital

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Losartan 50 mg / HCTZ 12.5 mg: Participants with mild to moderate essential hypertension who will receive Losartan 50 mg / Hydrochlorothiazide (HCTZ) 12.5 mg once-a-day for 12 weeks.
Period: Overall Study
Arm/Group | Losartan 50 mg / HCTZ 12.5 mg
Started | 15
Completed | 13
Not Completed | 2
Not completed — Lack of Efficacy | 1
Not completed — Unable to Follow Protocol Procedures | 1

BASELINE CHARACTERISTICS:
Arm/Group | Losartan 50 mg / HCTZ 12.5 mg
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Trough Sitting Diastolic Blood Pressure (SiDBP) at Week 12
Description: Participants with SiDBP of 95-115 mmHg at the end of Baseline had SiDBP measured after 12 weeks of treatment.
Time Frame: At Baseline and Week 12
Population: Intention-to-Treat
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Losartan 50 mg / HCTZ 12.5 mg
Number analyzed (Participants) | 15
mm Hg
  Baseline (N = 15) | 99.2 (5.5)
  Change from Baseline at Week 12 (N = 13) | -12.7 (3.2)
Statistical Analysis 1: Comparison: Losartan 50 mg / HCTZ 12.5 mg; Comparison of Week 12 and Baseline; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Losartan 50 mg/HCTZ 12.5 mg
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 8/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Losartan 50 mg/HCTZ 12.5 mg (N=15)
ARRHYTHMIA (Cardiac disorders) | 1 (1)
PALPITATIONS (Cardiac disorders) | 1 (1)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1)
BLOOD CHOLESTEROL INCREASED (Investigations) | 1 (1)
BLOOD GLUCOSE ABNORMAL (Investigations) | 2 (2)
BLOOD POTASSIUM DECREASED (Investigations) | 1 (1)
BLOOD SODIUM INCREASED (Investigations) | 1 (1)
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 2 (2)
BLOOD UREA INCREASED (Investigations) | 1 (1)
BLOOD URIC ACID INCREASED (Investigations) | 3 (3)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.